CLINICAL TRIAL: NCT01905514
Title: ImPRoving Adherence to Immunosuppressive Therapy by Mobile Internet Application in Solid Organ Transplant Patients
Acronym: PRIMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jongwon Ha, Professor of, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRIMA-13-002
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Kidney Transplantation

ARMS (2):
- control (No Intervention): using Medication event monitoring system
- internet mobile application (Active Comparator): using both mobile internet application and medication event monitoring system
  Interventions: Device: internet mobile application

INTERVENTIONS:
Device: internet mobile application
  Arms: internet mobile application

SUMMARY:
Nonadherence to immunosuppression is a leading cause of late graft rejection, chronic rejection and graft failure and it is regarded as a preventable cause of graft loss after solid organ transplantation. The purpose of this study is to evaluate whether mobile application for drug medication can enhance the drug adherence rate.

ELIGIBILITY:
Inclusion Criteria:

* 1 year after kidney transplantation
* out-patient follow up in Seoul National University Hospital
* using android smartphone
* taking Prograf as a main immunosuppressant
* 15-70 years

Exclusion Criteria:

* patients who cannot use medication event monitoring system
* multiorgan transplant
* immunosuppression medication change within 4 weeks of randomization
* caregiver management of the medication regimen
* pregnancy
* patients who can not use mobile application

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12-01 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
adherence rate | up to 6 months

SECONDARY OUTCOMES:
biopsy proven acute rejection rate | up to 6 months

OTHER OUTCOMES:
renal function | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jongwon Ha, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829